CLINICAL TRIAL: NCT06903078
Title: Pathogenic Exosomes During Herpes Zoster Mediate Increased Vascular Dementia Risk.
Brief Title: A Study That Collects Participant Data and Biospecimens to Analyze Pathogenic Exosomes That Mediate Increased Vascular Dementia Risk in Individuals With Herpes Zoster.
Acronym: R01
Status: Recruiting | Type: Observational
Sponsor: Center for Clinical Studies, Texas (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1R01AG085406-01 (NIH); R01AG085406 (NIH)
Record Dates: First submitted 2025-03-24; First posted 2025-03-30 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Herpes Zoster (HZ); Vascular Dementia
Keywords: RO1; 1R01AG085406-01; Herpes Zoster; Shingles; Dr. Stephen Tyring; Dementia risk HZ; VZV
MeSH Terms: conditions — Herpes Zoster; Dementia, Vascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample collection by venipuncture with butterfly needle collection kit; total blood volume collected at each visit is 20cc which is <2 Tablespoons of blood.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HZ (Herpes Zoster) Group: Participants with untreated acute herpes zoster outbreak.
- Control Group: Participants without acute herpes zoster outbreak.

SUMMARY:
The purpose of this observational research study is to study if patients with herpes zoster, also known as Shingles, have a higher risk of vascular dysfunction (problems with blood vessels, including stroke) and vascular dementia (problems with mental decline as a result of decreased blood flow to the brain) compared to patients without herpes zoster.

Patients are evaluated based on the group they are assigned too:

1. Herpes Zoster (HZ) Group: individuals presenting with untreated herpes zoster. These participants will have 6 visits:

   * Day 1 = 1st day presenting to clinic with acute zoster
   * 7 days post zoster
   * 1 month after Day 1
   * 3 months after Day 1
   * 6 months after Day 1
   * 12 months after Day 1
2. Control Group: individuals without herpes zoster o Day 1 (only 1 visit will be completed)

This study does not have a study medication/device. Standard of care for all patients will be followed.

DETAILED DESCRIPTION:
Vascular dementia: Vascular dementia is the second most common form of dementia after Alzheimer's disease and is characterized broadly as a loss of blood supply to the brain and compromised blood-brain barrier (BBB) ultimately leading to brain atrophy and cognitive impairment. Cerebrovascular insults such as stroke, myocardial infarctions, inflammation, and hyperactive platelets (thrombosis) are contributors and risk factors for the development of vascular dementia. Recently viruses have been identified as potential risk factors.

Varicella zoster virus (VZV) and vascular dysfunction: VZV is an exclusively human, double-stranded DNA alphaherpesvirus that produces varicella (chickenpox) then establishes latency within sensory and autonomic ganglionic neurons in >95% of adults in the U.S. With aging and immunosuppression, VZV reactivates in at least 1 in 3 individuals to produce herpes zoster (HZ; shingles) and other neurological diseases with or without rash. Despite the availability of two HZ vaccines, more than 1 million Americans develop HZ annually. Lesser known to the general public is the frequency of VZV reactivation without rash (zoster sine herpete). Given that VZV reactivates from ganglionic neurons across the entire neuraxis, essentially all organs and tissues, including the vasculature, are prone to infection and disease without the characteristic and diagnostic HZ rash. In fact, it is predicted that for every 1 case of HZ with rash, 7 individuals will reactivate with VZV without corresponding rash. Furthermore, the group has shown that individuals can still shed active virus in their saliva up to 12 years post-HZ suggesting at least a subset of individuals may have ongoing replication despite no rash; in this study 67% of patients still had active virus in their saliva at least 3 months post-rash. Thus, the burden of VZV disease, particularly duration, is likely grossly underestimated.

HZ is recognized as a stroke risk factor; HZ increases the risk of stroke up to 1 year post-HZ, with risk higher when HZ occurs in the ophthalmic distribution or in individuals <40 years of age. Specifically, data pooled from 9 studies in the U.S., Europe, and Asia show that the relative risk for stroke after HZ was 1.78 (95% CI 1.70-1.88) for the first month following HZ, dropping progressively to 1.20 (95% CI 1.14-1.26) after 1 year. Stroke risk increased by a larger margin during the first month after a HZ ophthalmicus episode: relative risk was 2.05 (95% CI 1.82-2.31); and the stroke risk remained elevated one year after the acute episode. A recent U.S. retrospective study of 23,339 HZ individuals and 46,378 controls, investigators found that during the 8 week aggregate period, HZ individuals were significantly more likely to suffer a stroke: adjusted incidence rate ratios for all patients and patients aged 18 to 49 years were 1.40 (95% CI, 0.93-2.11) and 8.12 (95% CI, 0.93-71.27), respectively (p < 0.05); risk returned to baseline by 1 year. The increased stroke risk in individuals with HZ who are < 50 years of age, compared to all HZ individuals, is remarkable because these individuals do not qualify for the HZ vaccine.

While the mechanisms underlying VZV and vascular disease are not fully elucidated, histological and immunohistochemical studies of VZV-infected arteries, analysis of cerebrospinal fluid (CSF) from VZV vasculopathy patients for cytokines and matrix metalloproteinases (MMPs), and in vitro studies provide some clues to the pathogenesis of disease (reviewed in Nagel and Bubak, 2018). Specifically, upon VZV reactivation, virus travels along nerve fibers that terminate in the outermost adventitial layer of the artery where virus-infected adventitial fibroblasts elicit a robust inflammatory response involving neutrophils early in disease, and T cells and macrophages throughout the entire course of disease. VZV-infected cells, neutrophils, and other infiltrating immune cells produce activated MMPs, which degrade the extracellular matrix potentially leading to weakening of the vessel wall, aneurysm formation, and rupture. Soluble factors secreted by inflammatory cells have also been described to further contribute to vascular smooth muscle death and accumulation of myofibroblasts in the thickened intima, potentially leading to arterial occlusion. However, the "soluble factors" have not been characterized until recently by the investigator group (described below).

Role of exosomes in disease states: Circulating exosomes have emerged as important "soluble factors" that can affect cells remote from their site of origin. Exosomes are small extracellular vesicles (~40-200 nm in diameter) of endosomal origin that carry cargo (proteins, nucleic acids, etc.) from their cells of origin to adjacent or distal cells for communication during normal and pathological states, regulating biological processes and response to disease. For example, exosomes derived from platelets, megakaryocytes, and peripheral blood mononuclear cells (PBMCs) can transfer CXCR4 and CCR5 to cells that lack these receptors, thereby increasing the number of susceptible cells for HIV infection. In other studies, exosomes released from nasopharyngeal carcinoma cells positive for EBV contain the viral latent membrane protein 1 and other viral/cellular factors that manipulate the tumor microenvironment to enhance tumor progression and alleviate immune responses to tumor cells. Furthermore, exosomes (and other extracellular vesicles) derived from:

1. breast cancer cells induce platelet activation and aggregation, contributing to cancer-associated thrombosis; and
2. VZV-infected primary human brain vascular adventitial fibroblasts mediate endothelial cell dysfunction and transmission of virions. The investigators have recently published a pilot study showing pathogenic plasma exosomes from patients with acute HZ are prothrombotic and proinflammatory. Specific proteins that were significantly elevated in HZ exosomes and involved in the platelet activation, signaling, and aggregation pathways included thrombospondin 1 (THBS1) caveolae-associated protein 2 (CAVIN-2), coagulation factor V (F5),56 and coagulation factor XIII A1 chain (F13A1)57 (Fig. 1). Cardiovascular system disease proteins elevated in HZ exosomes included calmodulin 1 (CALM1) and transthyretin (TTR) (Fig. 1). Elevated calmodulin 1 may contribute to oxidative stress associated with neural cell death after hypoxic-ischemic brain injury and is a predictor of poor stroke outcomes. Although increased serum transthyretin has been associated with improved ischemic stroke outcomes,60 transthyretin can also oligomerize and induce oxidative stress, inflammation and cell toxicity. Indeed, during HZ, amyloid-promoting factors are present in plasma, 8 potentially causing aggregation of increased circulating transthyretin to the toxic oligomeric form in arteries reminiscent of cerebral amyloid angiopathy (CAA).

Link between vascular dementia and VZV: As described above, VZV has been shown to be a causative agent of the aforementioned risk factors (stroke, vascular inflammation, etc.). Furthermore, a recent epidemiological study from two independent databases (FinnGen and UKB) found VZV reactivation significantly increases the risk of developing vascular dementia in particular (2.33 and 6.22, respectively; hazard ratios). A barrier in the acceptance of VZV and viruses in general to the development of vascular dementia and Alzheimer's disease is the lack or inconsistent presence of virus antigen/nucleic acids in the diseased tissues at time of death. While this can be potentially explained by a "hit-and-run" phenomenon (virus infects tissues, causes irreversible damage but is subsequently cleared), the investigators propose that non-infectious exosomes produced in the periphery (dorsal root and trigeminal ganglia) can contribute to disease distant from site of viral replication. The mechanisms in which VZV directly contributes to vascular dementia pathology in the absence of a lytic infection has not been studied and is the focus of this proposal. Taken together, the investigators hypothesize that circulating exosomes during HZ and in subsequent months will promote vasculitis and thrombosis, thus providing a mechanistic basis for the increased vascular dysfunction risk preceding vascular dementia.

SIGNIFICANCE: Strong epidemiological and correlational data exists linking VZV and dementia, including vascular disease and Alzheimer's disease. However, a paucity of mechanistic evidence has resulted in a hesitancy to causatively link the two. Thus, this proposal aims to address this gap in knowledge by systematically testing the role of pathogenic, long-lasting exosomes following HZ on vascular disease processes. Mechanistically uncovering proteins/miRNAs of interest can potentially change clinical practice with regards to duration of antiviral therapy and use of anti-platelet agents for HZ, as well as increase support for vaccination to prevent rash and mitigate stroke and vascular dementia risk. Furthermore, findings will serve as a model for how other pathogens can have long-lasting effects at sites remote from regions of infection and stimulate further research on the biological consequences of pathogen-associated exosomes.

INNOVATION AND IMPACT: This proposal has several areas of innovation. The longitudinal characterization and mechanistic investigation of circulating exosomes during HZ and 12-months post will:

1. provide a mechanistic understanding to the epidemiologically observed increased risk of vascular dementia and stroke following HZ. The direct contributions of viruses to dementia, including vascular dementia and Alzheimer's disease, is still controversial given most data linking the two are epidemiological and correlational. Data generated in this proposal will provide unbiased mechanistic information on how VZV can directly lead to vascular disease, contributing much-needed causative evidence of an early-stage risk factor or lack thereof.
2. change clinical management. Currently, modifiable stroke and vascular disease risk factors include hypertension, smoking, diabetes and hypercholesterolemia. Because these pathogenic exosomes increase risk of thrombosis and vasculitis, stroke risk factor modification should include HZ vaccination with the non-live subunit vaccine (Shingrix). If HZ occurs, longer duration antiviral therapy may be warranted as determined by results showing the length of time these pathogenic exosomes persist, as well as anti-platelet and anti- inflammatory agents. When available, there may also be a use for novel therapeutics that prevent exosome release/fusion.
3. change the paradigm of infectious disease. Typically, the investigators assume that once the clinical features of an infectious agent have resolved (such as rash from VZV reactivation), its subsequent impact on human health is negligible. The presence of pathogenic exosomes circulating for months in the absence of the triggering infectious agent suggests that clinicians need to consider infectious history remote from the time of stroke or vascular disease presentation.
4. employ new, cutting edge technology (ExoView R200) that will allow sorting and characterization of single exosomes to help us understand the population heterogeneity. These results, along with the larger body of results from the 2 Aims (including exosome sequencing data), will provide data for future grants to elucidate the function and cells of origin of the exosome subsets.

Study Rationale Aim 1. Analyze exosome content for known vascular damaging proteins/miRNAs from matched control and HZ individuals over a 12-month period. Using mass spectrometry and small RNA sequencing, the investigators will quantify abundance and temporal changes of exosomal proteins and miRNAs associated with vascular dysfunction, inflammation, coagulation, and stroke, then correlate analytes with clinical and laboratory features (anti-VZV IgG titers and IgM, complete blood counts, comprehensive metabolic panel, and aPTT/PT/INR). Enrichment analyses will be conducted on the network of exosomal proteins and miRNAs to uncover pathways and shared analytes associated with HZ, vascular dysfunction, and neurodegenerative processes.

Rationale: The investigators have recently published that during acute HZ, plasma exosomes contain elevated THBS1 and other proteins associated with vascular dysfunction. However, the longitudinal persistence of these risk factor proteins is not known and is imperative to uncovering the mechanisms mediating long-term vascular dementia risk and ultimately targeted interventional therapies beyond antiviral treatments. Given the epidemiological data correlating HZ reactivation and an increase in dementia diagnosis within 5 years, and more recently, the strong correlation of HZ reactivation and vascular dementia risk, the investigators predict certain risk factor proteins and miRNAs will remain elevated for up to a year following HZ reactivation. Temporal dynamics of the risk factor proteins are a critical step beyond acute timepoints because, typically, following rash clearance individuals are no longer on antiviral therapy, the extension of which could prove to be a clinically feasible and cost-effective way to reduce risk.

Aim 2. Determine the mechanism(s) in which non-infectious HZ exosomes promote vascular dysfunction. Plasma exosomes isolated from control and HZ individuals at timepoints above will be applied to human vascular endothelial cells derived from healthy donors or donors with APOE4 allele, then conditioned supernatant analyzed for proinflammatory cytokines (IFN-γ, IL-1β, IL-2, IL-4, IL-6, IL-8, IL-10, IL-12p70, IL-13, and TNF-α) by multiplex ELISA. Cells will also be analyzed for reactive oxygen species (ROS) generation and amyloid deposition. Additionally, the investigators will expose platelets from healthy donors to control and HZ exosomes to assess platelet function by quantification of: (1) platelet activation (upregulation of P-selectin, αIIbβ3, and phosphatidylserine) by flow cytometry; (2) platelet adhesion and aggregation in microfluidic flow assays; and (3) platelet retraction by clot contraction assays. The investigators will then correlate functional assay results with clinical and lab features (above), including the development of stroke and other vascular events in the individuals up to 12 months post-HZ. Knock-down experiments of specific proteins such as thrombospondin-1 will be conducted to investigate the mechanism of pathogenesis at the molecular level.

Rationale: The investigators propose to investigate the pathogenic effects of HZ exosomes on three cell types integral to vascular dementia, namely brain vascular adventitial fibroblasts (HBVAFs), vascular endothelial cells (VECs), and platelets. By doing so, the investigators aim to uncover the mechanisms underlying the epidemiological evidence of VZV- induced elevated risk of vascular dementia. Firstly, HBVAFs are known to play a key role in vascular disease and dysfunction, through the production of reactive oxygen species (ROS) and cytokines, as well as proliferation and migration of the adventitia during VZV vasculopathy cases.10 The preliminary study showed that HBVAFs exposed to HZ plasma exosomes taken at 3-months post-HZ induced the secretion of IL-6 and IL-8, which are key regulators of inflammation and vascular wall structure and function, compared to control plasma exosomes. However, the duration of this effect, other cytokines, and ROS production has not been elucidated, and could play a fundamental role in chronic vascular dysfunction seen in individuals up to 12 months post-HZ. Secondly, VECs are also key components in vascular dysfunction observed in vascular dementia cases, with an increase in ROS production and proinflammatory cytokine release, as well as a disruption in tight junctions mediating blood-brain-barrier integrity. Moreover, APOE4 allele carrying individuals are at an elevated risk of developing vascular dementia, as APOE4 expressing VECs exhibit a heightened proinflammatory and prothrombotic state compared to other APOE isoforms. Therefore, the investigators propose to investigate whether the pathogenic effects of HZ exosomes are exacerbated in APOE4 carrying individuals, by comparing VECs derived from both a carrier and non-carrier of APOE4. Lastly, vascular dementia is characterized by an occlusion of blood flow to the brain, with platelet hyperactivity observed in patients. The previous study revealed that HZ exosomes during acute HZ induced platelet activation and platelet-leukocyte aggregations. However, the duration of this effect is unknown and will be tested out to 12 months post-HZ, with and without clinically used anti-platelet agents. The finding of a long-lasting impact of HZ exosome on platelet activation and corresponding mitigating effect of anti-platelet drugs could represent a clinically feasible therapeutic intervention.

Previous reports have described a pro-inflammatory role for THBS1 in exosomes when exposed to macrophages. The pilot study and preliminary data shows a robust increase in THSB1 in exosomes of HZ patients but not controls.8 Therefore, to test whether the elevated load of THBS1 in HZ exosomes is responsible for the increase in cytokine release and ROS production, the investigators will conduct the HBVAF and VEC exposure experiments in the presence and absence of a THBS1 inhibitor, LSKL. Furthermore, THBS1 is a potent activator of TGFB1 and overproduction of TGFB1 is observed in Alzheimer's and vascular disease and induces cerebrovascular amyloidosis. Therefore, the THBS1 inhibitor will also be used in the amyloid deposition assays to evaluate exosome-carrying, THBS1-mediated amyloid formation in vascular cells.

STUDY DESIGN This study is a non-interventional/observational study that collects participant data and biospecimens in order to analyze exosome content for known vascular damaging proteins/miRNAs in HZ individuals over a 12 month period (6 visits) compared to control group (one visit).

Aim 1. Analyze exosome content for known vascular damaging proteins/miRNAs from matched control and HZ individuals over a 12-month period.

Anticipated results and interpretations: Based on preliminary and published pilot study results, the investigators expect to measure a significant increase in exosome proteins associated with thrombosis and vascular disease ("risk factor proteins") including THBS1, CAVIN-2, F5, F13A1, CALM1, and transthyretin (TTR) in plasma exosomes obtained from acute HZ individuals (initial visit) compared to those obtained from controls. Furthermore, the investigators expect these exosomal proteins in HZ individuals to remain at similar levels during the initial visit and 7 days later because patients would have been on antiviral therapy; then at 1 and 3 months, the investigators expect an increase in these proteins in a subset of individuals who still have ongoing viral replication that was merely slowed with antivirals; these individuals would have VZV IgG titers that did not decrease since the initial visit (decreasing VZV IgG titers are reflective of productive VZV infection resolving and virus returning to latency), rising VZV IgG titers since initial visit, or persistent VZV IgM or conversion of VZV IgM from negative to positive. In other words, the investigators predict that the VZV IgG levels will correspond to these elevations in the proteins of interest in a subset of HZ individuals, suggesting ongoing viral replication without rash in certain patients. Indeed, the group has previously reported the persistent shedding of VZV in the saliva of 67% of HZ individuals from 3 months to 12 years following HZ without the presence of a rash.56 Thus, the elevations of exosomal risk factor proteins in HZ individuals may be due to the incomplete shutdown of virus. The investigators expect these risk factor proteins to peak at approximately 3 months post-HZ, then decline at 6- and 12-months post-HZ because a study of VZV vasculopathy individuals showed the mean time from HZ to stroke is approximately 4 months.57 Additionally, given that the stroke risk is highest for individuals with HZO,10 the investigators expect exosomes from HZO individuals will have the highest level of risk factor proteins amongst all HZ individuals. As predicted in the preliminary studies, the investigators do not expect to find viral proteins or cytokines in the exosomes of control and HZ individuals.

With regards to RNA sequencing of HZ exosomes, the investigators do not expect to see any viral transcripts because VZV DNA and RNA is rarely detected during HZ (personal communications, Professor Ravi Mahalingam). The investigators expect to detect alterations in miRNAs implicated in cerebro- and cardiovascular disease such as miR-221 and miR-222 which are elevated in individuals with vascular disease, miR-143 which is an important mediator of pulmonary arterial hypertension, and miR-31 which increases oxidative stress in vascular smooth muscle cells. Interestingly, a preliminary study in the laboratory showed the significant elevation of these miRNAs in exosomes of VZV-infected sensory neurons compared to exosomes from mock infected neurons (Fig. 2). Finally, the investigators expect APOE4 carrying individuals to have the most robust and persistent risk factor proteins/miRNAs in their circulating exosomes given APOE4 is a known risk factor for vascular dementia.

Aim 2. Determine the mechanism(s) in which non-infectious HZ exosomes promote vascular dysfunction.

Anticipated results and interpretations: The pilot cytokine studies showed an increase in the production of IL- 6 and IL-8 from HBVAFs (which are key regulators of inflammation and vascular wall structure and function) following exposure to HZ exosomes compared to controls (Fig. 3). The investigators predict this will continue to be the case with a larger sample size and occur in the VECs. The investigators hypothesize these cytokines and ROS production will peak at the 1- and 3-month timepoints. For most individuals, the investigators hypothesize the ability to induce inflammation and ROS in naïve cells will diminish by 12-months post-HZ, however, APOE4 carrying VECs will likely remain hyper- inflammatory. The investigators have also conducted this assay using exosomes derived from mock- or VZV-infected human sensory neurons in vitro. Compared to mock exosomes, VZV-conditioned exosomes (which are non-infectious) applied to naïve HBVAFs significantly increased secretion of IL-6, IL-8, and IL-1β; therefore, the investigators suspect that the exosomes that trigger inflammatory cytokine production originate from VZV-infected cells. Given that the investigators see a prolonged elevation of HZ exosomes containing elevated risk factor proteins and these HZ exosomes can still induce IL-6 and IL-8 at 3 months post-HZ2 suggests there is ongoing viral replication in (a subset or all) HZ patients well after rash has cleared. As noted above, the group showed active VZV shedding in the saliva of HZ patients up to 12 years after clearance of rash. The investigators also predict to observe amyloid deposition in cells exposed to HZ exosomes but not controls and that this effect will be most prominent in the APOE4 carrying VECs. Finally, immunofluorescent staining will likely show a reduction in tight junction staining in HZ exposed VECs indicative of a disruption of blood-brain-barrier integrity. The investigators believe the pathogenic processes are due, in part, to the elevated load of THBS1 in HZ exosomes and that blocking the activity of THBS1 will attenuate these effects.

Based on the pilot study, the investigators anticipate seeing an increase in platelet activation as measured by an increase in platelets expressing P-selectin and phosphatidylserine following exposure to HZ exosomes but not control exosomes. Furthermore, the investigators predict this activation pattern will still be prominent at the 3-month time point indicative of a sustained risk for stroke, consistent with epidemiological data; the 20% exosome exposure from HZ samples is likely to have a more pronounced activation pattern than 10%. The investigators expect the activation pattern at 12 months post HZ will be diminished and not significantly different from control exosomes. Similarly, the investigators anticipate seeing an increase in rate and amount of platelet and fibrin accumulation in the microfluidic models of platelets exposed to HZ exosomes compared to platelets exposed to control exosomes. The investigators expect the CD36 inhibitor to attenuate the HZ exosome-induced effects on platelet function, which will provide strong mechanistic evidence. Using multiple methodologies to test platelet activation, aggregation, and function, as well as the induction of proinflammatory cytokine, ROS, and amyloid production by HBVAFs and VECs, the investigators will generate a comprehensive functional profile for HZ exosomes at various timepoints throughout disease. Results from these studies will have critical implications for clinical practice and how the investigators think of VZV reactivation in general. Specifically, if HZ exosomes are shown to be pathologically active and confer a functional increased risk of stroke and vascular dysfunction, as the preliminary data suggest, then longer antiviral treatment and/or anti-platelet therapies are warranted. Finally, it is likely the investigators will identify specific proteins in the exosomes via mass spectrometry (in Aim 1) that will correlate with the functional/mechanistic assays proposed in Aim 2. This could provide further therapeutic interventional targets and preliminary data for future knock-down experiments where exosomal proteins of interest are blocked to see if platelet activation is attenuated.

ELIGIBILITY:
Inclusion Criteria:

At the Screening Visit (Visit 1/Day 1), all participants must meet all the following criteria in order to be considered for participation in the study:

1. Be a male or female ≥ 18 years of age.
2. Present to clinic for routine dermatologic evaluation with or without rash.
3. Are willing and able to complete study visits and procedures, and able to effectively communicate with the investigator and other study personnel.
4. Have adequate venous access and are willing to undergo venipuncture for blood draws.
5. Able to provide written informed consent prior to any study procedures. Additional inclusion criteria for Herpes zoster (HZ) participants,
6. Present with acute, vesicle-stage HZ that has not been treated with antiviral therapies
7. Are willing and have reliable transportation to complete additional follow-up visits at 7 days, 1 month, 3 months, 6 months, and 12 months after initial visit for acute HZ.

Exclusion Criteria:

At the Screening Visit (Visit 1/Day 1), participants meeting any of the following criteria will be excluded from participation in the study:

1. Female individuals who are pregnant or breast-feeding.
2. Receiving systemic or topical antivirals for varicella zoster virus (VZV).
3. Sensitivity or allergy to systemic or topical antiviral medications for HZ.
4. History of diagnosed HZ within the last 8 years.
5. Received a HZ vaccine (e.g., Zostavax®/Shingrix®) within the last 8 years.
6. Received any vaccinations within the last 3 months.
7. Currently taking immunosuppressive therapies, including medications and radiation.
8. Currently taking any anticoagulants.
9. History of any coagulation disorder(s).
10. History of end-stage renal disease or uremia.
11. History of end-stage liver disease.
12. History of HIV.
13. Have had a COVID-19 infection in last 3 months.
14. Any history of non-skin cancers within the last 3 months.
15. History of serious infection requiring hospitalization in the last 3 months.
16. Prior history of cardiovascular accident or myocardial infarction within the last 12 months.
17. Prior cerebrovascular accident in the past 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Each year, 50 control subjects and 25 zoster individuals will be recruited to provide blood samples for this study, as well as clinical and laboratory information. This study will recruit individuals reflective of the United States demographics: 58% white (non-Hispanic), 19% Hispanic, 12% Black/African American, 6% Asian, and 5% two or more races. Houston is the fourth most populous city in the United States and has a demographic breakdown and population pool conducive to reflect the United States population. We will aim to recruit the following annually for years 1-5: (1) of the 50 control subjects, 29 White (non-Hispanic), 10 Hispanic, 6 Black/African American, 3 Asian, 2 Other (two or more), and (2) of the 25 control subjects, 14 White (non-Hispanic), 5 Hispanic, 3 Black/African American, 2 Asian, 1 Other (two or more). Within each ethnic group, half will be women and half men.
Sampling Method: Non-Probability Sample
Enrollment: 375 (Estimated)
Dates: Start 2025-02-13 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Analyze exosome content for known vascular damaging proteins/miRNAs from matched control and HZ individuals over a 12-month period. | From enrollment throughout the 5-year proposal period, occurring in a cyclical and overlapping manner.
  Using mass spectrometry and small RNA sequencing, we will quantify abundance and temporal changes of exosomal proteins and miRNAs associated with vascular dysfunction, inflammation, coagulation, and stroke, then correlate analytes with clinical and laboratory features (anti-VZV IgG titers and IgM, complete blood counts, comprehensive metabolic panel, and aPTT/PT/INR). Enrichment analyses will be conducted on the network of exosomal proteins and miRNAs to uncover pathways and shared analytes associated with HZ, vascular dysfunction, and neurodegenerative processes.

SECONDARY OUTCOMES:
Determine the mechanism(s) in which non-infectious HZ exosomes promote vascular dysfunction. | From enrollment throughout the 5-year proposal period, occurring in a cyclical and overlapping manner.

CONTACTS AND LOCATIONS:
Overall Officials: Project Director, Study Director — University of Colorado, Denver
Locations (2):
- United States (2):
  - Center for Clinical Studies, LTD. LLP, Houston, Texas
  - Center for Clinical Studies, LTD. LLP, Webster, Texas

IPD SHARING:
Plan to Share IPD: Yes
Direct identifiers such as name and initials will not be shared with those that conduct future research, unless required by law or patient safety. Personal Health Information may be shared with others for future research. Written authorization will be obtained from all participants in order to release this information to secondary researchers. All information shared with secondary researchers will be coded with the participant's PID, and every effort will be made to maintain the participant's confidentiality. Informed consent and HIPAA authorization will be obtained from all participants prior to collection of data and specimens. Those researchers involved in future research may receive medical history and study data, including demographics such as age, gender, race and ethnicity that are specific to the participant. Data and leftover samples will be coded and identified using a participant identification number (PID). Names and initials will not be shared.

REFERENCES:
- [Background] Richter ER, Dias JK, Gilbert JE 2nd, Atherton SS. Distribution of herpes simplex virus type 1 and varicella zoster virus in ganglia of the human head and neck. J Infect Dis. 2009 Dec 15;200(12):1901-6. doi: 10.1086/648474. PMID 19919304
- [Background] Nagel MA, Rempel A, Huntington J, Kim F, Choe A, Gilden D. Frequency and abundance of alphaherpesvirus DNA in human thoracic sympathetic ganglia. J Virol. 2014 Jul;88(14):8189-92. doi: 10.1128/JVI.01070-14. Epub 2014 Apr 30. PMID 24789785
- [Background] Mahalingam R, Wellish M, Wolf W, Dueland AN, Cohrs R, Vafai A, Gilden D. Latent varicella-zoster viral DNA in human trigeminal and thoracic ganglia. N Engl J Med. 1990 Sep 6;323(10):627-31. doi: 10.1056/NEJM199009063231002. PMID 2166914
- [Background] Gilden DH, Rozenman Y, Murray R, Devlin M, Vafai A. Detection of varicella-zoster virus nucleic acid in neurons of normal human thoracic ganglia. Ann Neurol. 1987 Sep;22(3):377-80. doi: 10.1002/ana.410220315. PMID 2823688
- [Background] Gershon AA, Chen J, Davis L, Krinsky C, Cowles R, Reichard R, Gershon M. Latency of varicella zoster virus in dorsal root, cranial, and enteric ganglia in vaccinated children. Trans Am Clin Climatol Assoc. 2012;123:17-33; discussion 33-5. PMID 23303966
- [Background] Iadecola C. The pathobiology of vascular dementia. Neuron. 2013 Nov 20;80(4):844-66. doi: 10.1016/j.neuron.2013.10.008. PMID 24267647